CLINICAL TRIAL: NCT02413372
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multiple Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamic Effects of BMS-986036 in Adults With Non-alcoholic Steatohepatitis
Brief Title: A Study of BMS-986036 in Subjects With Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB130-045
Record Dates: First submitted 2015-04-07; First posted 2015-04-09 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: First Line Therapy; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pegbelfermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group A: BMS-986036 (Experimental): Administered as specified on specified days
  Interventions: Drug: BMS-986036
- Treatment Group B: BMS-986036 (Experimental): Administered as specified on specified days
  Interventions: Drug: BMS-986036
- Treatment Group C: Placebo (Placebo Comparator): Administered as specified on specified days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-986036
  Arms: Treatment Group A: BMS-986036
Drug: BMS-986036
  Arms: Treatment Group B: BMS-986036
Drug: Placebo
  Arms: Treatment Group C: Placebo

SUMMARY:
The purpose of this study is to determine whether BMS-986036 is effective in the treatment of subjects with Non-alcoholic Steatohepatitis (NASH).

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male or female between 21 and 75 years old
* Body Mass Index (BMI) of 25 or more

Exclusion Criteria:

* Chronic Liver disease other than NASH
* Uncontrolled diabetes
* Any major surgery within 6 weeks of screening
* Unable to self-administer under the skin injections
* Any bone trauma, fracture or bone surgery within 8 weeks of screening

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (17):
  - Inland Empire Liver Foundation, Rialto, California
  - University Of California, San Diego, San Diego, California
  - Indiana University Health - University Hospital, Indianapolis, Indiana
  - Saint Louis University, St Louis, Missouri
  - Unc Hospitals And Clinics, Chapel Hill, North Carolina
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Upmc Center For Liver Diseases, Pittsburgh, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research PLLC, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - St. Luke'S Episcopal Hospital - Baylor College Of Medicine, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Sanyal A, Charles ED, Neuschwander-Tetri BA, Loomba R, Harrison SA, Abdelmalek MF, Lawitz EJ, Halegoua-DeMarzio D, Kundu S, Noviello S, Luo Y, Christian R. Pegbelfermin (BMS-986036), a PEGylated fibroblast growth factor 21 analogue, in patients with non-alcoholic steatohepatitis: a randomised, double-blind, placebo-controlled, phase 2a trial. Lancet. 2019 Dec 22;392(10165):2705-2717. doi: 10.1016/S0140-6736(18)31785-9. Epub 2018 Dec 13. PMID 30554783
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 184 participants enrolled; 80 entered lead-in phase; 75 were randomized and treated. Those did not enter lead-in phase: 95 no longer met study criteria; 5 withdrew consent; 1 poor/non-compliance; 3 other reasons. 2 from lead-in phase not randomized as no longer met study criteria. 3 from lead-in phase were randomized in the PK cohort (sub-study).
Groups:
- BMS-986036 10 mg QD: Participants self-administered 10 mg subcutaneous (SC) injections of BMS-986036, once daily (QD), for 16 weeks in a double-blind, outpatient setting.
- BMS-986036 20 mg QW: Participants self-administered 20 mg SC injections of BMS-986036, once weekly (QW), for 16 weeks in a double-blind, outpatient setting. The injection for days 2-7 of each treatment week was placebo to maintain the blind between daily and weekly treatment arms.
- Placebo QD: Participants self-administered SC injections of placebo, once daily, for 16 weeks in a double-blind, outpatient setting.
Period: Treatment
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Started | 25 | 24 | 26
Completed | 24 | 22 | 25
Not Completed | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Follow-up
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Started | 22 | 21 | 25
Completed | 20 | 20 | 23
Not Completed | 2 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Subject Withdrew Consent | 1 | 0 | 1
Not completed — Subject unable to return for visit | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD | Total
Number analyzed (Participants) | 25 | 24 | 26 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All treated participants
  years | 52.2 (9.99) | 51.5 (12.09) | 45.5 (11.89) | 49.7 (11.62)
Age, Customized [Count of Participants; unit: Participants] — Age categorization
  Participants
    < 65 years of age | 23 | 21 | 25 | 69
    >= 65 years of age | 2 | 3 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Female | 15 | 17 | 16 | 48
    Male | 10 | 7 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Hispanic or Latino | 7 | 6 | 7 | 20
    Not Hispanic or Latino | 18 | 18 | 19 | 55
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 1 | 0 | 1 | 2
    White | 24 | 23 | 25 | 72
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Hepatic Fat Fraction [Mean (Standard Deviation); unit: Percentage] — Population: All treated participants
  Percentage | 17.771 (7.2119) | 19.736 (5.8524) | 21.282 (7.3312) | 19.615 (6.9272)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Percent Hepatic Fat Fraction (%) by Magnetic Resonance Imaging (MRI) From Baseline to Week 16
Description: The mean change in percent hepatic fat fraction (%) by MRI from baseline to Week 16 was assessed for each arm. A longitudinal repeated measures analysis was used to analyze the change in hepatic fat fraction (%) at Week 16 from baseline in the treated population who have both a baseline and at least one post-baseline measurement.
Time Frame: From Day 1 to Day 112
Population: All treated participants
Measure: Mean (90% Confidence Interval); unit: percentage
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
percentage
  Day 57: number analyzed (Participants) | 24 | 21 | 24
  Day 57 | -8.43 [-9.81 to -7.06] | -6.45 [-7.90 to -5.00] | -1.26 [-2.58 to 0.06]
  Day 112: number analyzed (Participants) | 23 | 22 | 25
  Day 112 | -6.77 [-8.64 to -4.91] | -5.20 [-7.13 to -3.26] | -1.35 [-3.13 to 0.43]
Statistical Analysis 1: Comparison: BMS-986036 10 mg QD vs Placebo QD; Day 57; Test type: Superiority; Mean Difference (Final Values) = -7.17, 90% CI 2-sided [-9.09 to -5.26] — mean difference in adjusted change from baseline vs placebo
Statistical Analysis 2: Comparison: BMS-986036 20 mg QW vs Placebo QD; Day 57; Test type: Superiority; Mean Difference (Final Values) = -5.19, 90% CI 2-sided [-7.14 to -3.25] — mean difference in adjusted change from baseline vs placebo
Statistical Analysis 3: Comparison: BMS-986036 10 mg QD vs Placebo QD; Day 112; Test type: Superiority; p = 0.0004, t-test, 1 sided; Mean Difference (Final Values) = -5.43, 90% CI 2-sided [-8.01 to -2.84] — mean difference in adjusted change from baseline vs placebo
Statistical Analysis 4: Comparison: BMS-986036 20 mg QW vs Placebo QD; Day 112; Test type: Superiority; p = 0.0084, t-test, 1 sided; Mean Difference (Final Values) = -3.85, 90% CI 2-sided [-6.47 to -1.23] — mean difference in adjusted change from baseline vs placebo

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The number of participants with on-study AEs was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants | 18 | 13 | 15

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: The number of participants with on-study SAEs was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants | 1 | 0 | 1

4. Primary Outcome: Number of Participants With Injection Site Reactions
Description: The number of participants with on-study injection site reactions was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants
  Injection Site Bruising | 2 | 2 | 0
  Injection Site Erythema | 1 | 1 | 1
  Injection Site Reaction | 1 | 1 | 0
  Injection Site Pain | 0 | 0 | 1
  Injection Site Rash | 0 | 1 | 0
  Injection Site Swelling | 1 | 0 | 0

5. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Description: The number of participants with on-study AEs leading to discontinuation was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants | 0 | 0 | 0

6. Primary Outcome: Number of Deaths
Description: The number of deaths was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: The number of participants whose worst toxicity grade increased from baseline to grade 3 or 4 (Toxicity Scale: DAIDS Version 1.0) is reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants
  Alanine Aminotransferase (ALT) | 1 | 1 | 2
  Glucose, Fasting - high | 0 | 1 | 0

8. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: The number of participants with out-of-range vital signs noted during interim or final vital sign assessments was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants | 17 | 16 | 14

9. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: The number of participants with out-of-range ECG intervals observed during interim or final electrocardiogram assessments was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants
  PR > 200 msec | 2 | 1 | 2
  QRS > 120 msec | 1 | 0 | 3
  QT > 500 msec | 0 | 0 | 0
  QTcF > 450 msec | 2 | 2 | 1
  QT change from baseline > 30 msec | 5 | 6 | 5
  QTcF change from baseline > 30 msec | 6 | 2 | 3

10. Primary Outcome: Number of Participants With Physical Examination Abnormalities
Description: The number of participants with abnormalities observed during interim or final physical examination assessments is reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants | 11 | 9 | 12

11. Primary Outcome: Mean Percent Change From Baseline in Bone Mineral Density by Dual Energy X-Ray Absorptiometry (DXA)
Description: The mean percent change in bone mineral density from baseline to day 112 reported for each arm.
Time Frame: From Day 1 to Day 112
Population: All treated participants with DXA data at baseline and 6 months
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Percentage
  Femoral Neck: number analyzed (Participants) | 23 | 21 | 22
  Femoral Neck | -2.79 (4.329) | -1.08 (2.744) | -0.11 (2.749)
  Hip: number analyzed (Participants) | 23 | 21 | 22
  Hip | -0.91 (2.422) | -1.10 (1.549) | -0.93 (3.438)
  Spine: number analyzed (Participants) | 23 | 21 | 22
  Spine | -1.19 (2.658) | -1.21 (2.394) | -1.32 (3.203)
  Total Body Less Head: number analyzed (Participants) | 15 | 18 | 18
  Total Body Less Head | -0.43 (1.483) | -0.35 (1.529) | 0.10 (1.545)

12. Secondary Outcome: Geometric Mean of Trough Observed Plasma Concentration (Ctrough) of BMS-986036 at Day 112
Description: The observed serum concentration of BMS-986036 before the next dose is administered (pre-dose concentration) was assessed for both C-terminal intact and total molecule. Geometric means are presented for each arm.
Time Frame: From Day 1 to Day 112
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 20 | 21 | 26
ng/mL
  C-Terminal Intact | 162 (78.8) | 10.9 (113) | NA (NA) — Only reported for drug intervention arms.
  Total | 3250 (52.7) | 1130 (53.8) | NA (NA) — Only reported for drug intervention arms.

13. Secondary Outcome: Number of Participants With Positive Anti-BMS-986036 Antibody (ADA) Response at Day 142
Description: Participants were monitored for antibodies to study medication using a validated ADA homogenous bridge assay with BMS-986036 and electrochemical luminescence detection. The number of treated participants with positive Anti-BMS-986036 antibody titers up to Day 142 with regards to baseline was reported for each arm.
Time Frame: From Day 1 to Day 142
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants | 23 | 15 | 0

14. Secondary Outcome: Number of Participants With Positive Anti-FGF21 Antibody Response at Day 142
Description: Participants were monitored for antibodies to FGF21 using a validated homogenous bridge assay with Met-FGF21 (recombinant produced) and electrochemical luminescence detection. The number of treated participants with positive Anti-FGF21 antibody titers up to Day 142 with regards to baseline was reported for each arm.
Time Frame: From Day 1 to Day 142
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
Number analyzed (Participants) | 25 | 24 | 26
Participants | 23 | 15 | 0

ADVERSE EVENTS:
Time Frame: Non-serious adverse events after first dose of study medication and within 7 days of last dose and serious adverse events after first dose of study medication and within 30 days of last dose (approximately 4 months).
Arm/Group | BMS-986036 10 mg QD | BMS-986036 20 mg QW | Placebo QD
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/24 | 1/26
Other Adverse Events (participants affected / at risk) | 13/25 | 10/24 | 11/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986036 10 mg QD (N=25) | BMS-986036 20 mg QW (N=24) | Placebo QD (N=26)
Cellulitis (Infections and infestations) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986036 10 mg QD (N=25) | BMS-986036 20 mg QW (N=24) | Placebo QD (N=26)
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 2
Frequent bowel movements (Gastrointestinal disorders) | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 2
Fatigue (General disorders) | 1 | 0 | 5
Injection site bruising (General disorders) | 2 | 2 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 3 | 2
Increased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 2 | 3
Glycosuria (Renal and urinary disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-06-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT02413372/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT02413372/SAP_001.pdf